CLINICAL TRIAL: NCT04042610
Title: Office Worker Behavior and Health Study
Acronym: OWBHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: #5190289
Record Dates: First submitted 2019-07-30; First posted 2019-08-02 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Sedentary Behavior
Keywords: sitting time, Stand-Up, Amazfit
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups: intervention or control after informed consent is obtained. The intervention will be conducted for 8-weeks and consist of two components: education and electronic prompt to interrupt sitting time. Upon receiving the electronic prompt, the intervention group is encouraged to participate in 2 minutes of physical activity. Both groups will be provided an Amazfit BIP device to record and submit their step count during weeks: 1,2,4, 6 and 8.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: electronic prompt to interrupt sitting time (Experimental): The intervention will consist of two components: education and an electronic prompt via the iOS application Stand Up and notification through the Amzafit BIP device. The Stand-Up application will generate a prompt every hour during the workday to interrupt sitting time and encourage 2 minutes of physical activity. The intervention group participants will be given verbal and written educational materials on the health benefits of incorporating physical activity throughout their workday as well as the health risks of a sedentary lifestyle. Suggestions and demonstrations of physical activity will be given including but not limited to: use a restroom further away from their workstation, take a brief walk around the office, walk-in place, stretch. In addition, they will record their steps via the Amazfit BIP device and submit their daily step counts for weeks: 1,2,4, 6 and 8.
  Interventions: Behavioral: Electronic Prompt for Interrupting Sitting Time
- Control Group (No Intervention): The control group will be given an Amazfit BIP device to record their steps. They will submit their daily steps counts for weeks: 1,2,4, 6 and 8.

INTERVENTIONS:
Behavioral: Electronic Prompt for Interrupting Sitting Time — An electronic prompt via the IOS application Stand-Up will be given through the Amazfit BIP device to interrupt sitting time every hour during the office workers workday. The office worker will engage in 2 minutes of physical activity with each prompt.
  Arms: Intervention: electronic prompt to interrupt sitting time

SUMMARY:
This is a randomized intervention study to determine if electronic prompted interruptions in sitting time have an effect on job satisfaction, musculoskeletal complaints, and sitting time.

DETAILED DESCRIPTION:
A sedentary lifestyle has been deemed deleterious to health. It contributes to many chronic diseases and illnesses as well as an increase in all-cause mortality. The objective of this study is to investigate if electronic prompted interruptions in sitting time can reduce sedentary behavior at work as well as have an effect on job satisfaction, and musculoskeletal complaints. The participants will be randomly assigned to one of two groups, intervention (n=31) and control (n=31). Informed consent, demographic and socioeconomic data will be obtained from each participant. A questionnaire that includes three different scales will be administered before and after the 12-week intervention to all participants: Occupational Sitting and Physical Activity Questionnaire, Job Satisfaction Index, and Nordic Musculoskeletal Symptoms. Also, physical data will be measured: BMI, percent body fat and waist circumference. All participants will be provided with the Amazfit BIP device to track steps during work hours. The intervention group will receive a prompt every hour during their workday via an iOS application, Stand-Up, through the Amazfit BIP device. The prompt is to interrupt sitting time and encourage two-minutes of physical activity. The intervention group will receive examples of physical activity in addition to educational material on the health benefits of increasing physical activity in the workplace via verbal instruction and written materials. Data analysis will be conducted to determine if there is a difference in sitting time between the two groups over time using repeated-measures ANOVA. Independent samples t-tests will be used to compare job satisfaction and the physical biomarkers for obesity among the intervention and control groups. Chi-square will be used to analyze the reported musculoskeletal complaints between the two groups. If necessary, all analyses will be controlled for age, gender, race/ethnicity, and socioeconomic status.

ELIGIBILITY:
Inclusion Criteria:

In generally good health. Access to an IOS device for the duration of the study.

Exclusion Criteria:

Pregnancy. Use of activity equipment or devices in the workplace. Extreme exerciser: run marathons, participates in team or competitive sports/activities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-04-03 (Actual)

PRIMARY OUTCOMES:
Sitting Time | Change measure: baseline and 6 weeks
  Percent of time sitting in a typical workday
Activity in steps | Change measure: week 2 and 6 weeks
  The number of steps taken during their workday

SECONDARY OUTCOMES:
An Index of Job Satisfaction | Change measure: baseline and 8 weeks
  This index is by Brayfield and Rothe. There are eighteen questions which assess job satisfaction utilizing a 5-point Likert scale.
Musculoskeletal complaints questionnaire | Change measure: baseline and 8 weeks
  The questionnaire is also known as the Nordic Musculoskeletal Questionnaire. It uses Yes or No response to assess whether or not the participant has had musculoskeletal trouble in their neck, shoulders, upper back, elbows, wrists/hands, lower back, hips/thighs, knees, or ankles/feet over the past twelve months, if musculoskeletal problems have prevented normal function or working during the past twelve months, or if there has been musculoskeletal trouble during the past seven days.

CONTACTS AND LOCATIONS:
Overall Officials: Hildemar Dos Santos, MD, DrPH, Principal Investigator — Loma Linda University
Locations (1):
- La Sierra University, Riverside, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Becker I, Wallmann-Sperlich B, Rupp R, Bucksch J. [Workplace Interventions to Reduce Sedentary Behavior: A Systematic Review]. Gesundheitswesen. 2019 Aug;81(8-09):606-614. doi: 10.1055/s-0043-112746. Epub 2017 Nov 6. German. PMID 29108081
- [Background] Brayfield, A. H., & Rothe, H. F. (1951). An index of job satisfaction. Journal of Applied Psychology, 35(5), 307-311. doi:10.1037/h0055617
- [Background] Buman MP, Mullane SL, Toledo MJ, Rydell SA, Gaesser GA, Crespo NC, Hannan P, Feltes L, Vuong B, Pereira MA. An intervention to reduce sitting and increase light-intensity physical activity at work: Design and rationale of the 'Stand & Move at Work' group randomized trial. Contemp Clin Trials. 2017 Feb;53:11-19. doi: 10.1016/j.cct.2016.12.008. Epub 2016 Dec 7. PMID 27940181
- [Background] Chau JY, van der Ploeg HP, Merom D, Chey T, Bauman AE. Cross-sectional associations between occupational and leisure-time sitting, physical activity and obesity in working adults. Prev Med. 2012 Mar-Apr;54(3-4):195-200. doi: 10.1016/j.ypmed.2011.12.020. Epub 2011 Dec 28. PMID 22227284
- [Background] Church TS, Thomas DM, Tudor-Locke C, Katzmarzyk PT, Earnest CP, Rodarte RQ, Martin CK, Blair SN, Bouchard C. Trends over 5 decades in U.S. occupation-related physical activity and their associations with obesity. PLoS One. 2011;6(5):e19657. doi: 10.1371/journal.pone.0019657. Epub 2011 May 25. PMID 21647427
- [Background] Commissaris DACM, Huysmans MA, Mathiassen SE, Srinivasan D, Koppes LLJ, Hendriksen IJM. Interventions to reduce sedentary behavior and increase physical activity during productive work: a systematic review. Scand J Work Environ Health. 2016 May 1;42(3):181-191. doi: 10.5271/sjweh.3544. Epub 2015 Dec 18. PMID 26683116
- [Background] Crawford, J. O. (2007). The Nordic Musculoskeletal Questionnaire. Occupational Medicine, 57(4), 300-301. doi:10.1093/occmed/kqm036
- [Background] Daneshmandi H, Choobineh A, Ghaem H, Karimi M. Adverse Effects of Prolonged Sitting Behavior on the General Health of Office Workers. J Lifestyle Med. 2017 Jul;7(2):69-75. doi: 10.15280/jlm.2017.7.2.69. Epub 2017 Jul 31. PMID 29026727
- [Background] Duncan, M. D., Kazi, A., & Haslam, C. O. (2013/05/16/May 16-19, 2013). Sedentary behaviour at work: The impact on employee health.
- [Background] Dunstan DW, Howard B, Healy GN, Owen N. Too much sitting--a health hazard. Diabetes Res Clin Pract. 2012 Sep;97(3):368-76. doi: 10.1016/j.diabres.2012.05.020. Epub 2012 Jun 9. PMID 22682948
- [Background] Foley B, Engelen L, Gale J, Bauman A, Mackey M. Sedentary Behavior and Musculoskeletal Discomfort Are Reduced When Office Workers Trial an Activity-Based Work Environment. J Occup Environ Med. 2016 Sep;58(9):924-31. doi: 10.1097/JOM.0000000000000828. PMID 27454397
- [Background] Gibbs BB, Hergenroeder AL, Katzmarzyk PT, Lee IM, Jakicic JM. Definition, measurement, and health risks associated with sedentary behavior. Med Sci Sports Exerc. 2015 Jun;47(6):1295-300. doi: 10.1249/MSS.0000000000000517. PMID 25222816
- [Background] Gilson ND, Ng N, Pavey TG, Ryde GC, Straker L, Brown WJ. Project Energise: Using participatory approaches and real time computer prompts to reduce occupational sitting and increase work time physical activity in office workers. J Sci Med Sport. 2016 Nov;19(11):926-930. doi: 10.1016/j.jsams.2016.01.009. Epub 2016 Feb 18. PMID 26922132
- [Background] Healy GN, Eakin EG, Owen N, Lamontagne AD, Moodie M, Winkler EA, Fjeldsoe BS, Wiesner G, Willenberg L, Dunstan DW. A Cluster Randomized Controlled Trial to Reduce Office Workers' Sitting Time: Effect on Activity Outcomes. Med Sci Sports Exerc. 2016 Sep;48(9):1787-97. doi: 10.1249/MSS.0000000000000972. PMID 27526175
- [Background] Jancey J, Tye M, McGann S, Blackford K, Lee AH. Application of the Occupational Sitting and Physical Activity Questionnaire (OSPAQ) to office based workers. BMC Public Health. 2014 Jul 29;14:762. doi: 10.1186/1471-2458-14-762. PMID 25069528
- [Background] Ektor-Andersen J, Orbaek P, Isacsson SO; Malmo Shoulder-Neck Study Group. Behaviour-focused pain coping: consistency and convergence to work capability of the swedish version of the chronic pain coping inventory. J Rehabil Med. 2002 Jan;34(1):33-9. doi: 10.1080/165019702317242686. PMID 11900260
- [Background] Loghmani A, Golshiri P, Zamani A, Kheirmand M, Jafari N. Musculoskeletal symptoms and job satisfaction among office-workers: a cross-sectional study from Iran. Acta Med Acad. 2013;42(1):46-54. doi: 10.5644/ama2006-124.70. PMID 23735066
- [Background] McGuckin T, Sealey R, Barnett F. Planning for sedentary behaviour interventions: office workers' survey and focus group responses. Perspect Public Health. 2017 Nov;137(6):316-321. doi: 10.1177/1757913917698003. Epub 2017 Mar 25. PMID 28345430
- [Background] Parry S, Straker L, Gilson ND, Smith AJ. Participatory workplace interventions can reduce sedentary time for office workers--a randomised controlled trial. PLoS One. 2013 Nov 12;8(11):e78957. doi: 10.1371/journal.pone.0078957. eCollection 2013. PMID 24265734
- [Background] Proper KI, Singh AS, van Mechelen W, Chinapaw MJ. Sedentary behaviors and health outcomes among adults: a systematic review of prospective studies. Am J Prev Med. 2011 Feb;40(2):174-82. doi: 10.1016/j.amepre.2010.10.015. PMID 21238866
- [Background] Raynor HA, Bond DS, Freedson PS, Sisson SB. Sedentary behaviors, weight, and health and disease risks. J Obes. 2012;2012:852743. doi: 10.1155/2012/852743. Epub 2011 Dec 11. No abstract available. PMID 22187638
- [Background] Shrestha N, Kukkonen-Harjula KT, Verbeek JH, Ijaz S, Hermans V, Pedisic Z. Workplace interventions for reducing sitting at work. Cochrane Database Syst Rev. 2018 Jun 20;6(6):CD010912. doi: 10.1002/14651858.CD010912.pub4. PMID 29926475
- [Background] Thorp AA, Kingwell BA, Owen N, Dunstan DW. Breaking up workplace sitting time with intermittent standing bouts improves fatigue and musculoskeletal discomfort in overweight/obese office workers. Occup Environ Med. 2014 Nov;71(11):765-71. doi: 10.1136/oemed-2014-102348. Epub 2014 Aug 28. PMID 25168375
- [Background] Urda JL, Lynn JS, Gorman A, Larouere B. Effects of a Minimal Workplace Intervention to Reduce Sedentary Behaviors and Improve Perceived Wellness in Middle-Aged Women Office Workers. J Phys Act Health. 2016 Aug;13(8):838-44. doi: 10.1123/jpah.2015-0385. Epub 2016 Mar 21. PMID 26998705
- [Background] Valipour Noroozi, M., Hajibabaei, M., Saki, A., & Memari, Z. (2015). Prevalence of Musculoskeletal Disorders Among Office Workers. Jundishapur Journal of Health Sciencei, 7(1), e27157. doi:10.5812/jjhs.27157